CLINICAL TRIAL: NCT01734265
Title: Prospective, Open Uncontrolled Study to Evaluate the Safety of Depigoid With Two Pollen Combinations (Grasses/Olea and Grasses/Parietaria)2000DPP/ml in Patients With Allergic Rhinitis or Rhinoconjunctivitis With or Without Seasonal Asthma.
Brief Title: Safety Clinical Trial With Depigopid 50% Grasses/50% Olea Europaea(2000DPP/ml) or Depigoid 50% Grasses/50% Parietaria Judaica(2000DPP/ml).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6078-PG-PSC-193; 2012-001699-12 (EudraCT Number)
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2012-11

CONDITIONS: Allergy; Rhinitis; Rhinoconjunctivitis; Seasonal Asthma
MeSH Terms: conditions — Hypersensitivity; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depigoid 50% Grasses/50% Olea europaea (2000DPP/ml) (Experimental): Depigoid 50%Grasses/ 50% Olea europaea (2.000 DPP/ml) The administration regimen will consist of a rush build-up regimen: 0.2 ml followed by 0.3 ml after 30 minutes if no adverse events occur a second maintenance dose of 0,5 ml 4 weeks later.
  Interventions: Drug: Depigoid 50% Grasses/50% Olea europaea (2000DPP/ml)
- Depigoid 50% Grasses/50% Parietaria judaica (2000DPP/ml) (Experimental): Depigoid 50%Grasses/ 50% Parietaria judaica(2.000 DPP/ml) The administration regimen will consist of a rush build-up regimen: 0.2 ml followed by 0.3 ml after 30 minutes if no adverse events occur a second maintenance dose of 0,5 ml 4 weeks later.
  Interventions: Drug: Depigoid 50% Grasses/50% Parietaria judaica (2000DPP/ml)

INTERVENTIONS:
Drug: Depigoid 50% Grasses/50% Olea europaea (2000DPP/ml)
  Arms: Depigoid 50% Grasses/50% Olea europaea (2000DPP/ml)
Drug: Depigoid 50% Grasses/50% Parietaria judaica (2000DPP/ml)
  Arms: Depigoid 50% Grasses/50% Parietaria judaica (2000DPP/ml)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerance of a rush build up administration of Depigoid forte pollen and the first maintenance dose administered 4 weeks later.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerance of a rush build up administration of Depigoid forte pollen and the first maintenance dose administered 4 weeks later. The treatment period consists, thus, of 4 weeks.

Primary variable:

•Number of subjects [%] suffering at least one immediate or delayed systemic reaction of grade 2 or higher during the 4-weeks treatment period [grading according to the 2006 EAACI standards

ELIGIBILITY:
Inclusion Criteria:

* Subject has dated and signed the informed consent.
* Men and women between 18 and 60 years of age (both inclusive).
* Individuals suffering symptoms of allergic rhinoconjunctivitis or rhinitis during at least the preceding year, with or without allergic seasonal asthma caused by a clinically relevant sensitization to pollens (grasses AND P. judaica or O. europaea). Asthmatic patients can be included in the trial only if seasonal asthma is controlled with a medium daily dose minor or equal to 800 μg/day of budesonide or an equivalent or minor or equal to 400 μg/day of budesonide or an equivalent plus a long-acting- β2 agonist.
* Asthmatic patients must be stable within 3 months prior to Visit 1 and on an stable inhaled steroid dose within 6 weeks prior to visit 1 and throughout the study. FEV1 must be ≥ 80% of predicted value.
* The IgE-mediated sensitization must be demonstrated by the following:

medical history AND IgE specific CAP RAST ≥ 2 to the suspected relevant pollens (grass pollen AND Olea and/or Parietaria) AND a positive skin prick test to grass and Olea and/or Parietaria.

Exclusion Criteria:

* Any contraindication for treatment with allergen specific immunotherapy.
* Forced expiratory volume in 1 s (FEV1) or peak expiratory flow (PEF) value <80% of the predicted normal value.
* Clinically relevant allergy symptoms due to sensitization to perennial allergens (mites, molds, epithelia) or other seasonal pollen which might interfere with the safety of the IMP.
* Asthma requiring a dose > 800 μg/day of Budesonide or an equivalent, without long-lasting beta-2 agonists or requiring a dose > of 400 μg/day of Budesonide or an equivalent plus a long-acting-β2 agonist to reach asthma control, according to the Global Initiative for Asthma (GINA 2010)
* Patients with non controlled bronchial asthma within 3 months prior to Visit 1.
* Patients with asthma who have been treated with systemic steroids within 3 months prior to V1.
* Patients with hospital admission due to asthma exacerbations within 1 year prior to V1.
* Acute or chronic inflammatory or infectious diseases of the airways.
* Chronic structural diseases of the respiratory system (for example, emphysema or bronchiectasis).
* Immune system diseases, both autoimmune diseases and immunodeficiency.
* Any disease involving a contraindication for the use of adrenaline (for example, hyperthyroidism).
* Serious uncontrolled diseases involving a risk for the subjects participating in this study
* Malignant disease with activity in the last 5 years.
* Excessive consumption of alcohol, drugs or medication.
* Serious psychiatric, psychological or neurological disorders.
* Systemic or topical treatment with beta-blocker drugs 1 week before visit 2.
* Treatment with substances interfering with the immune system 2 weeks before visit 2.
* Use of tricyclic, tetracyclic and IMAO antidepressants. It will not be allowed to wash up antidepressants to enter the study because of the risks of interrupting antidepressant treatment, so patients on antidepressants therapy cannot be included in the trial.
* Use of systemic corticosteroids 3 months before visit 1.
* Immunization with prophylactic (bacterial or viral) vaccines within 7 days before visit 1 (prophylactic vaccines are allowed during the administration of IMP period provided they are administered at least one week after IMP administration and the next IMP administration is administered at least 14 days later).
* Participation of the subject in another clinical trial 30 days before visit 2
* Subjects who are going to donate stem cells, blood, organs or bone marrow in the course of the study.
* Female subjects who are pregnant or nursing and women with a positive pregnancy test at visit 1 or 2.
* Women of childbearing potential not using highly effective methods of birth control.
* Subjects who are unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
immediate or delayed systemic reaction of grade 2 or higher during the treatment period | 4 weeks
  The primary variable in this study is the number of subjects [%] who experienced at least one immediate or delayed systemic reaction of grade 2 or higher during the treatment period.

SECONDARY OUTCOMES:
immediate and/or delayed systemic reactions and immediate and/or delayed local reactions | 4 weeks
  Number of subjects [%] suffering immediate and/or delayed systemic reactions broken down by grade (EAACI classification).
  * Number of subjects [%] suffering immediate and/or delayed local reactions broken down by diameter (< 5 cm, 5-10 cm or > 10 cm).
  * Number of immediate and/or delayed systemic reactions broken down by grade (EAACI classification).
  * Number of immediate and/or delayed local reactions broken down by diameter (< 5 cm, 5-10 cm and > 10 cm).
  * (Immunology assessment):Measurement of the following immunological parameters: sIgE and sIgG4 at baseline and at the end of the study (after two maintenance doses).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Guardia, Dr, Principal Investigator — H. Virgen Macarena; Joaquín Quiralte, Dr, Principal Investigator — H. Virgen del Rocío; Luis Angel Navarro, Dr, Principal Investigator — H. Luis Alcañiz; Santiago Nevot, Dr, Principal Investigator — H. Manresa
Locations (4):
- Spain (4):
  - H. Manresa, Manresa, Barcelona
  - H. Virgen Macarena, Seville, Sevilla
  - H. Virgen del Rocío, Seville, Sevilla
  - H. Luis Alcañiz, Xàtiva, Valencia